CLINICAL TRIAL: NCT03143868
Title: Role of Acute Exercise Modality on Appetite Regulation and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16-2697; UL1TR001082-04 (NIH)
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Appetite Regulation; Acute Exercise; Energy Intake
Keywords: acute exercise; resistance exercise; aerobic exercise; appetite; energy intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise (Experimental)
  Interventions: Behavioral: Exercise Modality
- Resistance Exercise (Experimental)
  Interventions: Behavioral: Exercise Modality
- No Exercise (Placebo Comparator)
  Interventions: Behavioral: Exercise Modality

INTERVENTIONS:
Behavioral: Exercise Modality — The overall aim of this study is to compare how acute exercise modality (e.g. resistance exercise vs. aerobic exercise) differentially influence hormonal and behavioral indices of appetite regulation and ad libitum energy intake. Both conditions will also be compared to a non-exercise control condition.

SUMMARY:
This study plans to learn more about how type of exercise influences measures of appetite regulation. In this study, investigators will be evaluating a resistance exercise session (using weight machines and free weights) and an aerobic exercise session (using a treadmill). Participants will also complete a sedentary control condition.

A secondary purpose is to compare sex-based differences in appetite-indices in response to exercise. Therefore, the responses to aerobic and resistance exercise will also be compared between men and women.

ELIGIBILITY:
Inclusion Criteria:

* All ethnic groups and both genders
* Age: 18-55 yrs (changed in September 2018 because trial we are modeling enrollment criteria on [NCT02047721] changed age range, so we adjusted for this trial as well)
* BMI: 18.5-40 kg/m2 (changed in June 2018 from original range of 27-35 kg/m2 in order to improve recruitment. This is because recruitment within our prior BMI range had been slower than anticipated and potential participants that have expressed interest have screened out because of this. Given that we are still limiting enrollment criteria to adults who are inactive, it is likely that most will have body fat levels above normative standards, and therefore still be classified as having excess adiposity, even if their BMI is below 25 kg/m2. Furthermore, given the pilot nature of this work we believe it is important to complete the trial in a timely manner. We anticipate alterations to the enrollment criteria helping with this effort.)
* Weight stable within ±5% in the last 6 months
* Physically inactive (not meeting current physical activity guidelines, by self-report, no resistance training in previous 12-months)

Exclusion Criteria:

* History of cardiovascular disease (CVD), diabetes mellitus, uncontrolled hypertension (defined as: systolic blood pressure >160 mmHg or diastolic blood pressure >100mmHg, as measured during the screening visit with participants seated quietly, following established guidelines39), renal disease (e.g. chronic kidney disease, polycystic kidney disease, nephritis, etc.), hepatic disease (e.g. cirrhosis, liver failure, fatty liver, jaundice, etc.), untreated thyroid disease (e.g. Grave's disease, Hashimoto's disorder, goiters, thyroid cancers, etc.), or any other medical condition affecting weight or energy metabolism. Participants who are deemed ineligible based upon uncontrolled hypertension criteria will be referred to their primary care physicians for treatment. If this conditions become controlled they will be allowed to be re-evaluated for inclusion in the current trial.
* Symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Unable to exercise due to cardiac, pulmonary, neurologic or orthopedic reasons.
* Significant gastrointestinal disorders including: inflammatory bowel disease requiring treatment within the past year, chronic malabsorptive conditions, chronic diarrhea, or active gallbladder disease.
* Currently smoking and/or nicotine use within the past 6 months.
* Treatment with medications known to significantly affecting appetite, weight, energy metabolism, energy intake or energy expenditure in the last 6 months (e.g. systemic corticosteroids, appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants).
* Weight loss or weight gain of >5% in past 6 months.
* History of surgical procedure for weight loss at any time (e.g. gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve); history of extensive bowel resection for other reasons.
* Currently pregnant (confirmed via urine pregnancy test), lactating or less than 6 months post-partum.
* Self-report of alcohol or substance abuse within the past 12 months.
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder, or score >20 on the EATS-26. Participants with a score >20 on the EATS-26 will be referred to their primary care physician for further evaluation.
* Major psychiatric disorder (e.g. diagnosis of schizophrenia, bipolar disorder, or other psychotic disorders).
* Current severe depression or history of severe depression within the previous year (based on reported history, study physician examination findings, and/or a score >21 on the CES-D). Participants meeting any of these criteria will be referred to their primary care physician and/or the emergency department (based upon study physician determined level of severity).
* Significant food intolerances/allergies that cannot be accommodated by the CTRC Metabolic Kitchen.
* Currently participating in or planning to participate in any formal weight loss or physical activity programs or clinical trials.
* Other medical, psychiatric, or behavioral limitations that may interfere with participation (as determined by study physician).
* Unable or unwilling to undergo study procedures
* Women who are peri- or post-menopausal, or report irregular menstrual cycles.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Change in Ghrelin Area Under the Curve (AUC) | At baseline and every 30 minutes for 3 hours following a breakfast meal
  Concentration of ghrelin values, overtime for each arm of the study
Change in Peptide YY (PYY) AUC | At baseline and every 30 minutes for 3 hours following a breakfast meal
  Concentration of PYY values, overtime for each arm of the study
Change in GLP-1 AUC | At baseline and every 30 minutes for 3 hours following a breakfast meal
  Concentration of GLP-1 values, overtime for each arm of the study. Added in December 2017 following receipt of additional funding to add this measure)

SECONDARY OUTCOMES:
Change in Hunger AUC | At baseline and every 30 minutes for 3 hours following a breakfast meal
  Subjective indicator of hunger values, overtime for each arm of the study. Evaluated via 100 mm visual analogue scales
Change in Satiety AUC | At baseline and every 30 minutes for 3 hours following a breakfast meal
  Subjective indicator of satiety values, overtime for each arm of the study. Evaluated via 100 mm visual analogue scales
Change in Prospective Food Consumption AUC | At baseline and every 30 minutes for 3 hours following a breakfast meal
  Subjective indicator of prospective food consumption values, overtime for each arm of the study. Evaluated via 100 mm visual analogue scales
Change in Ad libitum Energy Intake - in lab | 3 hours following breakfast meal on each arm
  In lab ad libitum buffet lunch (via weigh and measure methodology) at the end of each study arm visit
Change in Ad libitum Energy Intake - free living | For 3 days following each arm
  3 days of free-living ad libitum energy intake (via self-report)

OTHER OUTCOMES:
Difference Between Men and Women in Appetite-Indices | At baseline, every 30 minutes for 3 hours following a breakfast meal, and for 3 days following each arm
  Sex-Based Differences (Added in December 2017 following receipt of additional funding to increase sample size for this purpose)
Difference in Behavioral Economics Constructs (Delayed Discounting and Hypothetical Purchase Task) | In the fed state, following completion of assigned exercise bout (or control bout).
  Delayed Discounting to evaluate value of future outcomes. Hypothetical Purchase Task to evaluate value of food. (Added in December 2017 following meeting with a colleague interested in adding these measures)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Halliday, PhD, RD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tobin SY, Cornier MA, White MH, Hild AK, Simonsen SE, Melanson EL, Halliday TM. The effects of acute exercise on appetite and energy intake in men and women. Physiol Behav. 2021 Nov 1;241:113562. doi: 10.1016/j.physbeh.2021.113562. Epub 2021 Sep 10. PMID 34516956
- [Derived] Halliday TM, White MH, Hild AK, Conroy MB, Melanson EL, Cornier MA. Appetite and Energy Intake Regulation in Response to Acute Exercise. Med Sci Sports Exerc. 2021 Oct 1;53(10):2173-2181. doi: 10.1249/MSS.0000000000002678. PMID 33831896